CLINICAL TRIAL: NCT02564705
Title: A Multi-Center, Prospective, Comparative Study of Anterior vs. Posterior Surgical Treatment for Lumbar Isthmic Spondylolisthesis
Brief Title: Comparative Study of Anterior vs. Posterior Surgical Treatment for Lumbar Isthmic Spondylolisthesis
Acronym: I-Spondy
Status: Completed | Type: Observational
Sponsor: AOSpine North America Research Network (Network)
Responsible Party: Sponsor
Other Study IDs: SPN-14-001
Record Dates: First submitted 2015-09-29; First posted 2015-10-01 (Estimated); Last update posted 2023-05-19 (Actual); Status verified 2023-05

CONDITIONS: Isthmic Spondylolisthesis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- anterior cohort: Anterior Lumbar Interbody Fusion (ALIF)
  Interventions: Procedure: Anterior Lumbar Interbody Fusion (ALIF)
- posterior cohort: * Posterolateral Fusion (PLF)
  * Posterior Lumbar Interbody Fusion (PLIF)
  * Transforaminal Lumbar Interbody Fusion (TLIF)
  Interventions: Procedure: Posterior Fusion

INTERVENTIONS:
Procedure: Anterior Lumbar Interbody Fusion (ALIF)
  Groups: anterior cohort
Procedure: Posterior Fusion — * Posterolateral Fusion (PLF)
  * Posterior Lumbar Interbody Fusion (PLIF)
  * Transforaminal Lumbar Interbody Fusion (TLIF)
  Groups: posterior cohort

SUMMARY:
The aim of this study is to compare outcomes and cost-effectiveness of anterior versus posterior surgical treatment for lumbar Isthmic Spondylolisthesis. The primary objective is to compare treatment effectiveness in terms of functional outcomes as measured by Oswestry Disability Index (ODI) v2.1a and to compare safety outcomes measured by treatment-related adverse events. Secondary objectives are to compare treatments in terms of differences in pain, quality of life, health utilities, and need for re-operation. Finally, a cost-effectiveness analysis will be performed. This analysis will take the form of cost-effectiveness if there is a difference in treatment effects or cost-minimization if there is no difference in treatment efficacy.

ELIGIBILITY:
Inclusion Criteria:

* Aged 18 to 80 years, inclusive
* Grade I, II or III (less than 75% slip of the cephalad vertebra compared to the caudal vertebra) isthmic spondylolisthesis at single level between L4 and S1
* Unresponsive to a minimum of 3 months of non-surgical treatment
* No previous surgical treatment for isthmic spondylolisthesis
* Patients who are medically suitable for surgical management
* Patients who have consented for surgical treatment
* Willing and able to comply with the Investigational Protocol (IP)
* Informed Consent Form (ICF) signed by patient

Exclusion Criteria:

* Any previous lumbar spine surgery
* Patient has significant scoliosis (Cobb angle is greater than 25 degrees)
* Subject has cauda equina syndrome defined as neural compression causing neurogenic bowel (rectal incontinence) or bladder (bladder retention or incontinence) dysfunction
* Subject is pregnant or of child-bearing potential and not currently on adequate birth control method
* Active infection at the surgical site
* Recent history (less than 1 year) of chemical substance dependency or significant psychosocial disturbance that may impact the outcome or study participation, in the opinion of the Investigator
* Pre-existent neurologic or mental disorder which would preclude accurate evaluation and follow-up (i.e. Alzheimer's disease, Parkinson's disease, unstable psychiatric disorder with hallucinations and/or delusions or schizophrenia
* Participation in another clinical trial of drug or device within the past 30 days that could influence the outcomes of this study
* Is a prisoner
* Acquired immune deficiency syndrome (AIDS) or AIDS-related complex
* Active malignancy or history of invasive malignancy within the last five years, with the exception of superficial basal cell carcinoma or squamous cell carcinoma of the skin that has been definitely treated; patients with carcinoma in situ of the uterine cervix treated definitely more than 1 year prior to enrollment may enter the study

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with Isthmic spondylolisthesis (IS)
Sampling Method: Non-Probability Sample
Enrollment: 177 (Actual)
Dates: Start 2016-03 (Actual); Primary Completion 2023-05-05 (Actual); Study Completion 2023-05-05 (Actual)

PRIMARY OUTCOMES:
Change in Oswestry Disability Index Score v2.1a | between pre-operative and 730 days (24 months)

SECONDARY OUTCOMES:
Change in Numeric Pain Rating Scale (Pain NRS) for low back pain | between pre-operative and 730 days (24 months)
Change in EQ-5D-3L health utility index | between pre-operative and 730 days

CONTACTS AND LOCATIONS:
Locations (14):
- United States (13):
  - University of California San Francisco, San Francisco, California
  - Carle Foundation Hospital, Urbana, Illinois
  - Kansas University Medical Center, Kansas City, Kansas
  - University of Maryland Medical Center, Baltimore, Maryland
  - Johns Hopkins University, Baltimore, Maryland
  - University of Missouri, Columbia, Missouri
  - Washington University, St Louis, Missouri
  - Cleveland Clinic, Cleveland, Ohio
  - Thomas Jefferson University / Rothman Institute, Philadelphia, Pennsylvania
  - Thomas Jefferson University, Philadelphia, Pennsylvania
  - University of Utah Department of Orthopedics, Salt Lake City, Utah
  - University of Virginia Department of Neurosurgery, Charlottesville, Virginia
  - Swedish Medical Center, Seattle, Washington
- Toronto Western Hospital, Toronto, Ontario, Canada